CLINICAL TRIAL: NCT06077604
Title: Influence of Air Pollution on SPondyloarthritis Flare-ups and Resistance to Treatment
Acronym: SPAIR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/811
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Spondyloarthritis, Axial
Keywords: Air pollution
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with a diagnosis of Axial Spondyloarthritis: Patients with a diagnosis of Axial Spondyloarthritis, received in rheumatology consultation/hospitalization over the period 2019-2022 and living in Franche-Comté over the same period
  Interventions: Other: Assessment of exposure to air pollution

INTERVENTIONS:
Other: Assessment of exposure to air pollution — For each patient, exposure to air pollution will be assessed over a period immediately prior to any flare-up and over four periods at a distance from the flare-up.

SUMMARY:
The relationship between exposure to air pollution and spondyloarthritis (SpA) has been poorly studied. Based on data from the literature on other inflammatory pathologies such as rheumatoid arthritis, we hypothesize that there is a relationship between exposure to air pollution and the risk of presenting a flare-up in SpA patients following and living in Franche-Comté (France).

Primary objective:The potential relationship between exposure to air pollution (nitrogen dioxide, fine particles with a diameter of less than 10 or 2.5 microns and Ozone) and the onset of a spondyloarthritis flare-up will be explored in patients with this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Axial Spondyloarthritis (radiographic or non-radiographic) according to Assessment of SpondyloArthritis international Society (ASAS) criteria
* Patient having received a consultation / hospitalization during the period 2019-2022
* Patient enrolled in the MISTIC cohort
* Having lived in Franche-Comté during the 2019-2022 period.

Exclusion Criteria:

* Other chronic inflammatory rheumatism (rheumatoid arthritis according to ACR 2010 criteria or psoriatic arthritis according to ClASsification criteria for Psoriatic ARthritis criteria)
* No inflammatory rheumatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Axial Spondyloarthritis, received in rheumatology consultation/hospitalization over the period 2019-2022 and living in Franche-Comté over the same period.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Occurrence of a SpA flare-up | 6 to 24 months
  The occurrence of a SpA flare-up measured by disease activity, defined according to the BASDAI (Bath Ankylosing Spondylitis Disease Activity Index) and/or ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score - C reactive protein) scores (BASDAI score ≥4/10 and/or ASDAS-CRP score ≥2.1) according to ASAS group

CONTACTS AND LOCATIONS:
Locations (1):
- Besançon University Hospital, Besançon, Bourgogne-Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No